CLINICAL TRIAL: NCT02682082
Title: A Randomize Double-Blind Control Trial Study Comparing Endoscopic Ultrasound-Guided Celiac Plexus Neurolysis W/Wo Bupivacaine In Patient Being Treated Palliatively For Pancreatic Cancer
Brief Title: EUS Guided Neurolysis Celiac Block w/wo Bupivacaine in Patient Being Treated Palliatively for Pancreatic Cancer
Acronym: EUS-CPN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by CHUM REB for incomplete documentation of research activities.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, A Sahai, Professeur Titulaire de Médecine / Professor of Medicine Chef / Chief, Service de Gastroentérologie, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CE 15.246
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Pain Management; Celiac plexus neurolysis; Bupivacaine; Palliative treatment
MeSH Terms: conditions — Pancreatic Neoplasms; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurolysis without Bupivacaine (Experimental): Experimental Group: Endoscopic ultrasound guided celiac plexus Neurolysis without Bupivacaine so only with Absolute Alcohol 20 mL
  Interventions: Procedure: Endoscopic ultrasound-guided celiax plexus neurolysis
- Neurolysis with Bupivacaine (Active Comparator): Endoscopic ultrasound guided celiac plexus Neurolysis with Bupivacaine (0.5% Bupivicaine 20mL + Absolute Alcohol 20 mL)
  Interventions: Procedure: Endoscopic ultrasound-guided celiax plexus neurolysis; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided celiax plexus neurolysis — Endoscopic ultrasound-guided celiax plexus neurolysis
Drug: Bupivacaine — Endoscopic ultrasound-guided celiax plexus neurolysis w/wo Bupivacaine
  Arms: Neurolysis with Bupivacaine

SUMMARY:
The goal of this project is to determine if EUS-CPN without Bupivacaine (versus EUS-CPN with Bupivacaine) can reduce pain scores and improve quality of life in patients with inoperable pancreatic cancer by reducing the morbidity due to narcotic side effects (e.g. nausea, excessive sedation, constipation).

DETAILED DESCRIPTION:
Pancreatic malignancies are the second highest incident gastrointestinal malignancy in Canada. From cancer mortality statistics in 2014, there were 4,700 new cases of pancreatic malignancies second only to colorectal cancer, representing 2.4% of all cancers . Even with chemotherapy, the median survival for patients with pancreatic adenocarcinoma is 6 to 10 months. Few of the patients are diagnosed at a resectable stage (12%-20%) so many patients are candidates for palliation only.In this context, one of the most important symptoms is pain because it often affects both quality of life and survival.70 to 80 % of patients with Pancreatic cancer had abdominal pain at the time of diagnosis . Adequate pain control is therefore an essential component of care in these patients. In the initial phase, the pain is visceral, but with disease progression, somatic pain may occur, especially due to the peripancreatic invasion of neural structures or muscles. Standard analgesics such as Acetaminophen are ineffective and administration of opioids is frequently limited by side effects such as nausea, constipation, somnolence, addiction, confusion or respiratory depression, and failure in achieving adequate analgesia. In these situations, neurodestructive methods of celiac plexus with Absolute Alcohol associated to Bupivacaine involving the main pancreatic pain pathways, seem efficient. Alcohol causes the immediate precipitation of endoneural lipoproteins and mucoproteins within the celiac plexus, leading to the extraction of cholesterol and phospholipids from the neural membrane. To prevent severe transient pain after the procedure, Bupivacaine was injected before the Alcohol injection. Interest and importance of EUS-CPN is well established (safe, more effective than percutaneous or CT guided celiac plexus Neurolysis, significant reduction in pain and significant reduction of narcotics requirements) however the role and effect of Bupivacaine on the effectiveness of Neurolysis and lytic power of Alcohol has never been studied . Is it a synergistic effect ? Or an antagonistic effect by diluting Alcohol ? The Centre hospitalier de l'université de Montréal (CHUM) is currently the busiest EUS center in the world and has the largest experience with EUS-guided CPN. The CHUM also probably see more pancreatic cancers annually than any other center (more than 300 proven cases/year). There are no published reports of serious adverse events associated with this procedure and this has been the investigators experience as well. Patients may however experience some mild to moderate discomfort during the initial injection of the absolute ethanol solution, but this is usually short lived (less than 30 minutes in our experience). Therefore, Bupivacaine is currently injected before the Ethanol injection, however, local anesthetic was not used before the Phenol injection for example because it has been reported that Phenol has an immediate local anesthetic effect.

The investigators believe that, Bupivacaine has no effect and instead it dilutes the alcohol and then reduces the lytic power of Ethanol. This study was designed to test this hypothesis prospectively.

The goal of this project is to determine if EUS-CPN without Bupivacaine (versus EUS-CPN with Bupivacaine) can reduce pain scores and improve quality of life in patients with inoperable pancreatic cancer by reducing the morbidity due to narcotic side effects (e.g. nausea, excessive sedation, constipation).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed malignant pancreatic lesion involving the pancreatic genu, body, or tail
* Abdominal or back pain considered to be potentially related to the tumor

  * New onset pain (<3 months)
  * Constant
  * Centrally located
  * With or without irradiation to the back
  * No obvious other source of pain based on history and physical examination by the attending endosonographer
* No possibility of surgical management
* Signed, informed consent

Exclusion Criteria:

* Allergy to bupivicaine
* Age < 18 years
* Inability or unwillingness to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Difference in pain scores at 1 month and end of the trial | 1 month and 120 days post procedure

SECONDARY OUTCOMES:
Difference in quality of life scores at 1 month and end of the trial | 1 month and 120 days post procedure
  Quality of life will be measured using the DDQ 15 quality of life instrument (a validated 15-question instrument specific for diseases of the digestive system)
Difference in cumulative narcotic usage at 1 month and end of the trial | 1 month and 120 days post procedure
Difference in survival | 1 month and 120 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anand Sahai, M.D, Principal Investigator — Hopital Saint Luc (Centre Hopitalier de l´Université du Montreal)
Locations (1):
- CHUM, Montreal, Quebec, Canada

REFERENCES:
- [Background] Seicean A. Celiac plexus neurolysis in pancreatic cancer: the endoscopic ultrasound approach. World J Gastroenterol. 2014 Jan 7;20(1):110-7. doi: 10.3748/wjg.v20.i1.110. PMID 24415863
- [Background] Wyse JM, Chen YI, Sahai AV. Celiac plexus neurolysis in the management of unresectable pancreatic cancer: when and how? World J Gastroenterol. 2014 Mar 7;20(9):2186-92. doi: 10.3748/wjg.v20.i9.2186. PMID 24605017
- [Background] Seicean A, Cainap C, Gulei I, Tantau M, Seicean R. Pain palliation by endoscopic ultrasound-guided celiac plexus neurolysis in patients with unresectable pancreatic cancer. J Gastrointestin Liver Dis. 2013 Mar;22(1):59-64. PMID 23539392
- [Background] Levy MJ, Chari ST, Wiersema MJ. Endoscopic ultrasound-guided celiac neurolysis. Gastrointest Endosc Clin N Am. 2012 Apr;22(2):231-47, viii. doi: 10.1016/j.giec.2012.04.003. Epub 2012 Apr 25. PMID 22632946
- [Background] Sakamoto H, Kitano M, Komaki T, Imai H, Kamata K, Kudo M. Endoscopic ultrasound-guided neurolysis in pancreatic cancer. Pancreatology. 2011;11 Suppl 2:52-8. doi: 10.1159/000323513. Epub 2011 Apr 5. PMID 21471704
- [Background] Penman ID. Coeliac plexus neurolysis. Best Pract Res Clin Gastroenterol. 2009;23(5):761-6. doi: 10.1016/j.bpg.2009.05.003. PMID 19744638
- [Background] Ishiwatari H, Hayashi T, Yoshida M, Ono M, Masuko H, Sato T, Miyanishi K, Sato Y, Takimoto R, Kobune M, Miyamoto A, Sonoda T, Kato J. Phenol-based endoscopic ultrasound-guided celiac plexus neurolysis for East Asian alcohol-intolerant upper gastrointestinal cancer patients: a pilot study. World J Gastroenterol. 2014 Aug 14;20(30):10512-7. doi: 10.3748/wjg.v20.i30.10512. PMID 25132769